CLINICAL TRIAL: NCT02750059
Title: Adjunctive Therapy With Telmisartan Instituted With ART During Acute HIV Infection to Reduce the Establishment of CNS Reservoirs of HIV and Lymph Node Fibrosis
Brief Title: Using Telmisartan With ART During Acute HIV Infection to Reduce the CNS Reservoirs of HIV and Lymph Node Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nittaya Phanuphak, MD, PhD, Nittaya Phanuphak, MD, PhD, SEARCH Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEARCH 018; 1R01NS084911-01 (NIH)
Record Dates: First submitted 2015-05-30; First posted 2016-04-25 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acute HIV Infection; HIV CNS Involvement
MeSH Terms: interventions — Telmisartan; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TDF/3TC/EFV + Telmisartan (Experimental): The subjects will receive 40mg telmisartan daily for 4 weeks followed by 80mg telmisartan daily for 44 weeks in addition to ART
  Interventions: Drug: TDF/3TC/EFV + Telmisartan
- TDF/3TC/EFV only (Active Comparator): Subjects will receive ART only
  Interventions: Drug: TDF/3TC/EFV only

INTERVENTIONS:
Drug: TDF/3TC/EFV + Telmisartan — The subject will receive 40mg telmisartan daily for 4 weeks followed by 80mg telmisartan daily for 44 weeks in addition to ART. Subjects unable to tolerate 80mg of telmisartan will be able to de-escalate to 40mg daily
  Other Names: tenofovir/lamivudine/efavirenz + Micardis
  Arms: TDF/3TC/EFV + Telmisartan
Drug: TDF/3TC/EFV only — Starting from the first visit, all participants will be placed on an ART regimen to treat HIV. This is the standard route of care for HIV patients.
  Other Names: tenofovir/lamivudine/efavirenz
  Arms: TDF/3TC/EFV only

SUMMARY:
Primary objective: To compare telmisartan therapy + antiretroviral therapy (ART) versus ART alone during acute Human Immunodeficiency Virus (HIV)a infection in reducing systemic immune activation and trafficking of activated and HIV-infected cells to the central nervous system (CNS), and limiting establishment and persistence of the CNS reservoir of HIV.

At 48 weeks (during the telmisartan therapy) and 72 weeks (~6 months after cessation of telmisartan augmentation), the investigator expect subjects in the telmisartan group will have reduced levels of blood and CSF immune activation markers, reduced brain inflammation, lower CSF HIV ribonecleic acid (RNA) and improved neuropsychological testing performance.

Secondary objective: In subjects who are willing to undergo the optional inguinal lymph node biopsy, the study will determine whether subjects receiving telmisartan plus ART for 48 weeks develop less lymphoid tissue fibrosis than subjects receiving ART alone for 48 weeks.

Subject population: Male and female subjects age ≥ 18 years old with acute HIV infection who are identified and enrolled in SEARCH 010/RV254 protocol will be asked to co-enroll in this study.

Number of subjects: 21

Duration of follow-up: 72 weeks

Study design: 21 acutely HIV-infected subjects will be randomized 2:1 to treatment with telmisartan + ART (n=14) vs. ART alone (n=7) for the first 48 weeks followed by ART alone in both arms to week 72. Blood and CSF, magnetic resonance imaging (MRI), and neuropsychological testing and exam will be collected at baseline, week 48 and week 72. Inguinal lymph node biopsy is an optional procedure that will be offered at baseline and week 48.

DETAILED DESCRIPTION:
Clinical assessments:

Neurological exam: South East Asia Research Collaboration with Hawaii (SEARCH) employs the AIDS Clinical Trials Group (ACTG)-derived HIV macroneurological examination, a physician rated symptoms assessment of cognitive features typical of HAND and peripheral neuropathy

Neuropsychological assessments: SEARCH employs the HIV neurocognitive battery originally developed by Maj et al. designed to minimize cultural bias and tested in Bangkok. All subjects will have the full SEARCH battery as previously published, avoiding evaluations following invasive procedures.

Quantification of Drug use: Drug and alcohol use are assessed with a structured interview including methamphetamine, heroin, and marijuana based on a Thai Red Cross study defining frequently abused drugs in Bangkok. Urine is stored at each visit and may be later tested for illicit drugs. Evidence of intoxication is documented so that neuropsychological data can be censored.

Lumbar punctures are completed per standard clinical procedures using a Sprotte® (pencil-point) needle to minimize complications. Standard assessments of CSF and serum, protein and cell count are completed and approximately 20cc are collected and ultra-centrifuged, Cell pellets of both blood and CSF will be cryopreserved for future potential studies, with subject consent. Supernatants are divided into 0.5cc aliquots, and frozen to -80oC on the same day. Venereal Disease Research Laboratory test (VDRL)/Rapid Plasma Reagin (RPR) will be assessed at baseline and in follow up if risk for new syphilis exposure is reported. Participant hospitalization for hydration will be completed, if needed. Participants will be compensated for their time based on Institutional Review Board (IRB)-approved rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Have protocol-defined acute HIV-1 infection (Tested 4th generation HIV enzyme immunoassay [EIA] negative and NAT positive or tested 4th generation HIV EIA positive, negative by less sensitive EIA and nucleic acid testing [NAT] positive)
3. Be part of the SEARCH 010/RV 254 study
4. Ability and willingness to start ART immediately after diagnosis
5. Understand the study and sign informed consent form. Persons who cannot read will have the consent form read to them by a member of the study staff and may then give informed consent by using making a thumb print
6. Availability for follow-up for the duration of the planned study
7. Systolic blood pressure ≥ 110 mmHg
8. Agree to undergo lumbar puncture at weeks 0, 48 and 72
9. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Pregnancy (current or within the last 6 months) or breastfeeding
2. Uncontrolled hypertension
3. Use of thiazolidinediones or other angiotensin receptor blockers class [losartan, irbesartan, olmesartan, valsartan, candesartan (washout permitted)]
4. Screening laboratory values: absolute neutrophil count (ANC) < 750 cells/mm3, hemoglobin <10 gm/dL creatinine clearance<30mL/min (estimated by the Cockcroft-Gault equation using ideal body weight)
5. Known renal artery stenosis
6. Known cirrhosis or severe liver disease
7. Unstable coronary artery disease/angina or decompensated congestive heart failure
8. Any history of intolerance to any angiotensin II receptor blocker (ARB)
9. Need for ongoing potassium supplementation
10. Any contraindication to lumbar puncture such as history of bleeding diathesis or known cerebral mass lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Difference between study arms at weeks 48 and 72 in CSF neopterin | 48 and 72 weeks

SECONDARY OUTCOMES:
Difference between study arms in lymphoid tissue fibrosis at week 48 | 48 weeks
Difference between study arms at weeks 48 and 72 in brain inflammation by magnetic resonance spectroscopy (MRS) | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in CSF HIV RNA by single copy assay | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in aggregate neuropsychological testing performance score (NPZ-4) on Grooved Pegboard, Color Trails 1, Color Trails 2 and Trail Making A | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in CSF monocyte chemoattractant protein-1 (MCP-1) levels | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in CSF interferon-gamma-inducible protein-10 (IP-10) levels | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in plasma neopterin levels | 72 weeks
Difference between study arms at weeks 48 and 72 in plasma soluable CD14 (sCD14) levels | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in plasma interleukin-6 (IL-6) levels | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in plasma D-dimer levels | 48 and 72 weeks
Difference between study arms at weeks 48 and 72 in plasma soluable CD163 (sCD163) levels | 48 and 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- SEARCH Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided